CLINICAL TRIAL: NCT06352229
Title: The Playful Learning in Infancy Program (PLIP): A Pilot Feasibility Study of an Universal Educational Parenting Program Using a Parallel Group Design
Brief Title: The Playful Learning in Infancy Program
Acronym: PLIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: LEGO Foundation (Unknown)
Responsible Party: Principal Investigator, Mette Væver, PhD, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 514-0335/23-2000
Record Dates: First submitted 2024-03-20; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Parent-Child Relations; Infant Development
Keywords: Universal intervention; Playful Learning; Infant; Parental competence; Socioemotional; Public health visitors; Prevention
MeSH Terms: interventions — Postnatal Care

STUDY DESIGN:
Intervention Model Description: Evaluation is based on a parallel group study, with half of the participants receiving care as usual and half of the participants receiving care as usual along with the Playful Learning in Infancy Program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Playful Learning in Infancy Program (Experimental): Playful Learning in Infancy Program plus postnatal care as usual
  Interventions: Behavioral: Playful Learning in Infancy Program
- Care As Usual (Active Comparator): Postnatal care as usual
  Interventions: Behavioral: Postnatal care as usual

INTERVENTIONS:
Behavioral: Playful Learning in Infancy Program — Research-based knowledge on play with babies delivered to the parents systematically by public health visitors based on a manual, activity cards, and video clips at four time points from 0 to 12 months postpartum.
  Other Names: Leg og samspil; Playful Interactions
  Arms: Playful Learning in Infancy Program
Behavioral: Postnatal care as usual — In accordance with Danish national guidelines, health visitors visit families during the infants first year of life, where they weigh and measure the infant. Further, they offer individual guidance and support regarding for instance feeding, sleeping, how to stimulate the infant, and the developmental stages that the infant goes through.
  Arms: Care As Usual

SUMMARY:
In the Playful Learning in Infancy Program, parents receive research-based educational guidance on playful interactions with their infants aged 0-1 year. They learn to recognize their infants' cues indicating readiness to engage in play and they are introduced to specific, developmentally appropriate activities for interactive engagement. The guidance is delivered to parents during routine home visits by public health visitors.

The aims of the Playful Learning in Infancy Program are to 1) promote playful interactions between infants and parents, parental attitudes towards play, and infant socioemotional development; 2) enhance the language and knowledge of playful learning in infancy among frontline staff; and 3) evaluate the Playful Learning in Infancy Program for potential testing in a future large-scale RCT study.

Evaluation is based on a parallel group study design, with half of the participants receiving care as usual and half of the participants receiving care as usual along with the Playful Learning in Infancy Program.

ELIGIBILITY:
Inclusion Criteria:

* Residence address in the Danish municipalities of Hvidovre or Billund
* Residence address with child or legal custody of the child
* Child is between 1-7 months old
* Understands Danish or English

Exclusion Criteria:

* Parental age under the age of 18 when the child is born
* Multiple pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2327 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Parental Playful interactions | T2 (infant age 3-3.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 10-10.5 months)
  Playful interactions are assessed using The Parent Play Questionnaire (PPQ) by Ahmadzadeh et al. (2020), which assesses the frequency of parent-child play and screen use.

SECONDARY OUTCOMES:
Parental Stress | T3 (infant age 7-7.5 months)
  Maternal and paternal parenting stress is assessed via self-report using the Parenting Stress Index™, Third Edition Short Form (PSI-3-SF; Abidin, 1995).
Infant Socio-emotional Development | T5 (infant age 11-11.5 months)
  Infant socio-emotional development is assessed via parental report using the Ages & Stages Questionnaires®: Social-Emotional, Second Edition (ASQ:SE-2; Squires, Bricker, & Twombly, 2015).
Infant Level of Play | T4 (infant age 10-10.5 months)
  We have developed questions for the parents to report on the child's level of play, based on Belsky, J., & Most, R. K. (1981).
Parental Mind-Mindedness | T5 (infant age 11-11.5 months)
  Parental mind-mindedness is assessed using a written response to the first question from the "Describe your child" interview (Meins et al., 1998). Mind-mindedness is coded according to the criteria specified in the mind-mindedness coding manual (Meins & Fernyhough, 2015).
Parental Attachment Style | T1/Enrollment (4 weeks - 8 months)
  Parents' attachment style is assessed using the Experience in Close Relationships-Revised-Short Form (ECR-RS) questionnaire (Fraley et al., 2000).
Parental Mental Well-Being | T1/Enrollment (4 weeks - 8 months) and T5 (infant age 11-11.5 months)
  Parental mental well-being is assessed using the Warwick-Edinburgh Mental Well-being Scale - (S)WEMWBS (Tennant et al., 2007).
Infant Screen Time | T2 (infant age 3-3.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 10-10.5 months)
  The infant's screen time is assessed using quantitative questions developed for the project and administered to parents.
Questions developed for the study regarding Parental Involvement | T2 (infant age 3-3.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 10-10.5 months)
  Questions developed for the study regarding the parent's involvement in the child's life and daily activities.
Questions developed for the study regarding Parental Knowledge of Play | T2 (infant age 3-3.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 10-10.5 months)
  Questions developed for the study for parents in the intervention group regarding knowledge of play.
Parental Experience of the PLIP | Immediately after the intervention
  Qualitative interviews with a subsample of parents.
Health Visitors' Experience of the PLIP | Immediately after the intervention
  Qualitative interviews with a subsample of health visitors.

CONTACTS AND LOCATIONS:
Overall Officials: Mette S. Væver, Principal Investigator — University of Copenhagen
Locations (1):
- Center for Early Interventions and Family Studies, Department of Psychology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No